CLINICAL TRIAL: NCT03681834
Title: Multi-center Register for the Use of the Cor-Knot® Automated Knotting System in Heart Valve Surgery
Acronym: RECORVA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MORGANT 2018
Record Dates: First submitted 2018-08-28; First posted 2018-09-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Vascular Surgery
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Data on the effectiveness and safety of the Cor-Knot® knotting device

SUMMARY:
The Cor-Knot® device is an automated knotting system for valve sutures and prosthetic rings used for more than a year during valve replacements and annuloplasties in cardiac surgery. It reduces the time spent knotting the threads fixing the prosthesis and thus reduces aortic clamping and extracorporeal circulation times. The originality of the project is based on the absence of national multi-rate data collection on the effectiveness and safety of the Cor-Knot® knotting device.

ELIGIBILITY:
Inclusion Criteria:

* programmed minimally invasive surgery for:

  * aortic valve replacement
  * mitral valve replacement
  * mitral valve plastic surgery
* adult patient

Exclusion Criteria:

* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring valve surgery
Sampling Method: Non-Probability Sample
Enrollment: 557 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Presence of periprosthetic leak around the prosthetic rings as determined during physical examination (rated yes/no ) | Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Morgant MC, Malapert G, Petrosyan A, Pujos C, Jazayeri S, Bouchot O. Comparison of automated fastener device Cor-Knot versus manually-tied knot in minimally-invasive isolated aortic valve replacement surgery. J Cardiovasc Surg (Torino). 2020 Feb;61(1):123-128. doi: 10.23736/S0021-9509.19.10792-6. Epub 2019 Oct 4. PMID 31599141